CLINICAL TRIAL: NCT00222716
Title: Improving Adherence to Antiretroviral Therapy
Brief Title: Managing Medications
Acronym: MM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Judith Erlen, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2R01NR004749 (NIH)
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: HIV Infections
Keywords: Treatment adherence; HIV; Self-efficacy; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Structured (Experimental): Behavioral Intervention: Structured counseling behavioral intervention focused on problem solving.
  Interventions: Behavioral: Problem solving counseling
- Usual Care (No Intervention): Control arm
- Inidividualized (Experimental): Behavioral Intervention: Individualized nurse counseling behavioral intervention focused on problem-solving
  Interventions: Behavioral: Problem solving counseling

INTERVENTIONS:
Behavioral: Problem solving counseling — Telephone nurse counseling behavioral intervention focused on problem solving.
  Arms: Inidividualized; Structured

SUMMARY:
The primary aim of this study is to compare the effect of an individualized adherence intervention (TI) and a structured adherence intervention (TS) to usual care on adherence to antiretroviral therapy in persons infected with HIV (PWHIV).

DETAILED DESCRIPTION:
The primary aim of this study is to compare the effect of an individualized adherence intervention (TI) and a structured adherence intervention (TS) to usual care on adherence to antiretroviral therapy in persons infected with HIV (PWHIV). The secondary aims address the relationship between adherence and quality of life (QOL), and between adherence and clinical response. The exploratory aims focus on examining the effect of self-efficacy on the relationship between the intervention and adherence, the effect of adherence on the relationship between self-efficacy and outcomes (clinical response and quality of life), as well as the effects of symptoms, alcohol and/or drug use, chronic interpersonal problems, mood, social support, optimism, perceived burden of medication regimen, perceived stigma, purpose in life, co-morbidity, personality, literacy, and intimate partner abuse on self-efficacy, and psychometric analyses of the instruments. The sample of 300 (plus 51 dropouts) PWHIV who are taking antiretroviral therapy and without cognitive dysfunction will be randomly assigned to one of two treatment arms. Those individuals who are deemed to be 100% adherers (approximately 25-50) will be assigned to the control group, but will be followed separately as a natural history substudy and interviewed. Data will be collected at baseline, post-treatment, post-maintenance, post-booster, and 18 months. Electronic event monitors, diaries, the Self-reported Medication-taking Scale, and the ACTG Adherence Follow-up Questionnaire will be used to assess adherence. The Digit Vigilance Test will be used to assess the effect of sustained attention on adherence. QOL will be measured using the MOS-HIV, the Satisfaction with Life Scale, and the Perception of Illness Visual Analogue Scale. Clinical response will be assessed using viral load, CD4 T-cell count, AIDS defining conditions, and hospitalizations. Variables influencing self-efficacy (measured with an investigator-developed Self-efficacy Scale) will be examined: symptoms ( CRCD Symptom Checklist), alcohol and/or drug use (AUDIT), chronic interpersonal problems (IIP), social support (Interpersonal Support Evaluation List), optimism (Life Orientation Test), anxiety (Beck Anxiety Inventory) and Beck Depression Inventory II), perceived burden of regimen (visual analog scales), perceived stigma (Perceived Stigma of HIV Scale), purpose in life (Purpose in Life Scale), co-morbidity (CRCD Co-Morbidity Scale), personality characteristics (NEO-FFI), health literacy (Test of Functional Health Literacy in Adults), knowledge about HIV medication adherence (HIV Medication Adherence Knowledge), and intimate partner abuse (Abuse Assessment Screen). A repeated measures model with planned comparisons will be used to test the hypotheses for the primary aim. Structural equation modeling will be used to examine the relationships identified in the secondary and exploratory aims. PWHIV who adhere to their therapy may live longer, require fewer hospitalizations, and have an improved QOL.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to give informed consent,
* be 18 years or older,
* be taking antiretroviral therapy,
* be able to speak and understand English,
* have a telephone or access to a telephone,
* and be living in a private residence or apartment in the community as opposed to a personal care/nursing home.

Exclusion Criteria:

* significant cognitive impairment,
* blind
* motor impairment of their upper extremities
* if another person in their household was or is currently enrolled in the study
* the HDS that we will use to screen for cognitive impairment cannot be used with individuals who have these physical problems
* Those with a hearing impairment who do not have a modified telephone to enhance their hearing will be excluded since they are unable to participate in the telephone delivered interventions or data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2004-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Medication adherence as measured by electronic event monitors | 12 weeks
  MEMS data using AARDEX medication monitoring caps, percent daily dose correct.

SECONDARY OUTCOMES:
Morisky Medication Adherence Scaler | 12 weeks
  9 item Morisky self report measure on medication adherence

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Erlen, PHD, Principal Investigator — University of Pittsburgh; Lisa K Tamres, MS, Study Director — University of Pittsburgh School of Nursing
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is not plan to share data specifically but the data has been shared with the Mach14 Collaborative. Entire data set has been shared with the Collaborative.

REFERENCES:
- [Derived] Butler KR, Harrell FR, Rahim-Williams B, Robinson JM, Zhang X, Gyamfi A, Erlen JA, Henderson WA. Symptoms and Comorbidities Differ Based on Race and Weight Status in Persons with HIV in the Northern United States: a Cross-Sectional Study. J Racial Ethn Health Disparities. 2023 Apr;10(2):826-833. doi: 10.1007/s40615-022-01271-0. Epub 2022 Mar 10. PMID 35274279